CLINICAL TRIAL: NCT03620435
Title: A Phase II Trial of Transurethral Surgery Followed by a Combination of Atezolizumab (Tecentriq™) an Anti-PDL-1 (MPDL3280A) With Trimodal Therapy in Patients With Muscle-Invasive Bladder Cancer
Brief Title: Trimodal Therapy Plus Atezolizumab in Muscle-invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Wassim Kassouf, Principle Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML-39576
Record Dates: First submitted 2018-07-23; First posted 2018-08-08 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Safety Issues
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- atezolizumab (Experimental): Atezolizumab will be given during trimodal therapy, and every 3 weeks for 16 cycles or until disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab (1200mg iv, every 3 weeks) administered concurrently with TMT and adjuvant for up to one year
  Other Names: Tecentriq

SUMMARY:
This is a single arm phase II trial to (1) evaluate safety and toxicity profile of intravenous Atezolizumab (anti-PDL-1) administered in combination with TMT in patients with MIBC, (2) To determine the loco-regional control rate (LCR) of TMT combined with PDL-1 blockade.

DETAILED DESCRIPTION:
This will be a Phase II trial (stage 1 and 2). This study will initially accrue 3 evaluable patients to assess the dose limiting toxicity (DLT) of combination of Gemcitabine (4 weeks at 100 mg/m2, given intravenously once weekly, 2-4 hours before radiation therapy) plus IMRT (50 Gy/20 fractions. 2.5 Gy per fraction - 5 times per week for 4 weeks) and Atezolizumab (1200 mg intravenous on day 1 of 3 week cycle. Once the first 3 patients are accrued, the trial will be placed on hold for 3 months until acute toxicity has been assessed and the combination is felt to be safe according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE,v. 4.03). DLT will be defined as: (1) Grade 3 or higher immune related Adverse Events (irAEs), (e.g. inflammatory ocular toxicities, pneumonitis, hepatitis, colitis), (2) Grade 3 or higher treatment-related AEs (TRAE) that delay EBRT by > 21 days. For the safety run-in component of the study, 3 patients will receive Atezolizumab at a dose of 1200 mg every 3 weeks, as described above. After the third patient has been accrued, the trial will be placed on hold for 3 months for an assessment of acute toxicity. Acute toxicity is defined as any toxicity occurring within 90 days from the end of the combined treatment of IMRT and gemcitabine. If no grade 3 or higher acute toxicity is detected, Atezolizumab 1200 mg will be chosen for the rest of the trial. If one patient develops grade 3 toxicity, 3 further patients will be entered at 1200 mg. . If no further grade 3 toxicity is observed, this dose level will be considered safe. In case that one additional patient develop a grade 3 toxicity, then 3 patients will be enrolled at the reduced dose of 840mg. If no grade 3 or higher acute toxicity is detected, Atezolizumab 840mg will be chosen for the rest of the trial. If one patient develops grade 3 toxicity at the reduced dose, then 3 further patients will be entered at 840 mg. If no further grade 3 toxicity is observed, this reduced dose level will be considered safe. In case that one additional patient develop a grade 3 toxicity at the reduced dose level, it will be considered too toxic and the combination will be judged too toxic for the population and regimen, and the study will be terminated.

If treatment is well tolerated, this will be considered the final dose for the study. No further de-escalation beyond this level will be considered. For the Stage 2 of this study,, up to 22 other patients will be accrued (total of 25 evaluable patients). Atezolizumab will be given during combination treatment, and every 3 weeks for 16 cycles or until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria

* 18 years old or older
* Histologic diagnosis of urothelial carcinoma of the bladder. Focal differentiation allowed other than small cell histology.
* Stage T2-T4a N0M0 (AJCC-TNM version 6) based on trans-urethral resection of bladder tumor (TURBT), CT imaging, +/- bimanual examination under anaesthesia (EUA).
* CT scan of chest/abdomen/pelvis within 8 weeks from the start of treatments, showing no evidence of metastatic disease.
* Attempt of complete TURBT within 56 days (8 weeks) prior to the start of chemoradiation. If TURBT was performed > 8 weeks ago but a recent cystoscopy show no residual disease, then a repeat TURBT is not necessary.
* Life Expectancy greater than 6 months
* ECOG performance status of 2 or better
* Another primary cancer is allowed only if treated with curative intent at least 3 years prior to enrollment without evidence of recurrence or if the untreated cancer is clinical indolent (eg lower risk prostate cancer).
* Adequate hematologic reserve: Platelet count ≥ 150,000/ul, WBC ≥ 4000/ul. Anemia will be corrected to minimum hemoglobin of 100 g/L with red cell transfusions, if necessary.
* Adequate liver function with a bilirubin ≤ 1.5 ULN[27] and SGOT/SGPT < 1.5 X the upper normal limit
* Patients must be considered able to tolerate systemic chemosensitizer combined with pelvic IMRT by the joint agreement of the participating radiation oncologist and medical oncologist.
* Able and willing to give written informed consent.

Exclusion criteria

* Prior systemic therapy for other urothelial tumors. Neoadjuvant chemotherapy can be considered a component of the trimodal therapy and is allowed. Superficial bladder treatments including BCG and mitomycin C are permitted if completed 6 weeks prior to therapy.
* Hypersensitive to Gemcitabine or to any ingredient in the formulation or component of the container.
* Prior RT to the pelvis
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days or five half-lives of the drug, whichever is longer, prior to enrollment
* Malignancies other than urothelial cancer within 5 years prior to Cycle 1, Day 1:

Patients with localized lower risk prostate cancer (defined as Stage ≤T2b, Gleason score ≤ 7, and PSA at prostate cancer diagnosis ≤ 20 ng/mL[if measured]) treated with radical prostatectomy and without prostate-specific antigen (PSA) recurrence are eligible.

Patients with lower risk prostate cancer (defined as Stage T1/T2a, Gleason score ≤ 7 and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.

Patients with malignancies of a negligible risk of metastasis or death (e.g., risk of metastasis or death <5% at 5 years) are eligible provided they meet all of the following criteria:

Malignancy treated with expected curative intent (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated surgically with curative intent) No evidence of recurrence or metastasis by follow-up imaging and any disease-specific tumor markers

* Pre-existing medical conditions precluding treatment (e.g. previous history of immune-related adverse reactions, pneumonitis, colitis, etc.)
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study. Patients with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
* Active tuberculosis
* Pregnancy or lactating mothers. Women of childbearing age must use contraception during treatment and for 5 months after the last dose of Atezolizumab. Acceptable methods are: oral contraceptives, hormonal implants, hormonal patches, IDU, Diaphragm with spermicides, cervical cape with spermicide, and condom with spermicide.
* Received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial
* Active autoimmune disease that has required systemic treatment in past 2 years
* Received or will receive a live vaccine within 4 weeks prior to first dose of study drug. Influenza vaccination should be given during influenza season only (approximately October through May in the Northern Hemisphere and approximately April through September in the Southern Hemisphere). Patients must agree not to receive live, attenuated influenza vaccine (e.g., FluMist®) within 28 days prior to randomization, during treatment or within 5 months following the last dose of atezolizumab (for patients randomized to atezolizumab)
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Serum albumin < 2.5 g/dL
* Active infection requiring IV systemic therapy
* Receipt of therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study
* Prior allogeneic stem cell or solid organ transplant
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Patients with active Hepatitis B virus (HBV) or Hepatitis C virus (HCV)
* Not willing or unable to sign a consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety profile of intravenous Atezolizumab (anti-PDL-1) administered in combination with TMT in patients with MIBC | 2-2.5 years
  Safety will be captured as (1) number of patients with Grade 3 or higher immune related Adverse Events (irAEs), (e.g. inflammatory ocular toxicities, pneumonitis, hepatitis, colitis), (2) number of patients with Grade 3 or higher treatment-related AEs (TRAE) that delay EBRT by > 21 days. The safety assessments up to the final follow-up visits will consist of monitoring and recording adverse events, including serious adverse events and adverse events of special interest, protocol-specified safety laboratory assessments, protocol-specified vital signs, and other protocol-specified tests that are deemed critical to the safety evaluation of the study.

SECONDARY OUTCOMES:
Overall survival | 4 years
  OS is defined as the time from start of treatment to date of death due to any cause. Patients who have not died at the time of the analyses cutoff / end of study, will be censored at their last contact date known to be alive). Patient will be followed for 3 years from completion of radiotherapy
Bladder cancer therapy impact on quality of life | 2-2.5 years
  Changes from baseline quality of life will be measured longitudinally using the validated Functional Assessment of Cancer Therapy-Bladder questionnaire. FACT-BL scores on the first day of chemo radiotherapy treatment (before starting treatment), on the week 3 of radiation therapy, and again at 3, 6, 12, 18, and 24 months post radiation therapy. Quality of life domains measured includes domains of physical well-being, social and family well-being, emotional well-being, and functional well-being, as well as additional concerns specific to patients undergoing therapy for bladder cancer such as urinary, bowel and sexual function.
Complete response to TMT combined with PDL-1 blockade | 2-2.5 years
  LCR (loco-regional control rate) or early complete response rates from the combined therapy is the proportion of patients with a confirmed locoregional complete response at 3 months post-radiation. Loco regional complete response will be ascertained on basis of a combination of follow-up CT imaging of the irradiated field (bladder, pelvic lymph nodes), cystoscopy with rebiopsy of involved areas, and urine cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Kassouf, MD, Study Chair — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- MUHC, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
no plan formulated yet